CLINICAL TRIAL: NCT03214887
Title: Therapeutic Angiogenesis for Peripheral Artery Occlusive Disease Using Hyaluronan Combined With Autologous Bone Marrow Cell Therapy -- Phase I/II Safety and Efficacy Study
Brief Title: Autologous BMMNC Combined With HA Therapy for PAOD
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Incomplete enrollment process
Sponsor: Academia Sinica, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AS-IRB-BM-14056
Record Dates: First submitted 2017-07-05; First posted 2017-07-12 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Peripheral Arterial Occlusive Disease; Critical Limb Ischemia
Keywords: Hyaluronan; Bone marrow mononuclear cells
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Intervention Model Description: RV-P1501-4: Gel-like product with 10 thousand BMMNCs in each ml of 1% hyaluronan (HA) solution
  RV-P1501-5: Gel-like product with 100 thousand BMMNCs in each ml of 1% hyaluronan (HA) solution
  RV-P1501-6: Gel-like product with 1 million BMMNCs in each ml of 1% hyaluronan (HA) solution
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RV-P1501-4 (Experimental): Gel-like product with 10 thousand BMMNCs in each ml of 1% hyaluronan (HA) solution
  Interventions: Biological: RV-P1501
- RV-P1501-5 (Experimental): Gel-like product with 100 thousand BMMNCs in each ml of 1% hyaluronan (HA) solution
  Interventions: Biological: RV-P1501
- RV-P1501-6 (Experimental): Gel-like product with 1 million BMMNCs in each ml of 1% hyaluronan (HA) solution
  Interventions: Biological: RV-P1501

INTERVENTIONS:
Biological: RV-P1501 — Gel-like product with BMMNCs in each ml of hyaluronan (HA) solution

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of hyaluronan combined with autologous bone marrow mononuclear cells for the treatment of critical PAOD patients.

DETAILED DESCRIPTION:
This is a multicenter, non-blinded and randomized study to evaluate the safety and efficacy of hyaluronan (HA) combined with autologous bone marrow mononuclear cells (BMMNC) therapy for critical peripheral arterial occlusive disease (PAOD) patients.

A total of 30 subjects will be recruited into the study. The subjects will be randomized into 3 different arms. During the Phase I study, 9 subjects recruited while another 21 additional subjects will be recruited in Phase II after the review of DSMB and consultation of Taiwan FDA on the results of the Phase I study.

Each subject will be administered 5~10 injections of RV-P1501, the number of injections depends on the size of the subject's ischemic leg. Each subject will receive treatment once. Subjects will be assigned to the treatments in random order. Evaluations including ABI, PWT/PFWT, clinical status, EF, CTA, biochemistry and hematology checked during the inclusion and exclusion evaluation, and will be taken at baseline, 1 week, 2 weeks, 4 weeks, 12 weeks, and 24 weeks after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 20
* Patients with severe PAOD and diagnosed with Rutherford category 3, 4, or 5
* Contraindication to angioplasty or bypass surgery, or post-angioplasty or bypass surgery for once but with limited or no effect.
* Patient without hypertension or hypertensive patient with adequate-controlled blood pressure.
* With signed informed consent

Exclusion Criteria:

* Patient undergone any organ transplantation
* Inability to undergo bone marrow aspiration
* Pregnant woman
* Life expectancy < 1 year
* Cognitive impairment
* Active malignancy in 5 years prior to treatment
* Bleeding diathesis or pulmonary embolism
* Patient with active major cardiovascular diseases such as unstable angina, arrhythmia, heart failure, impaired cardiac function (ejection fraction < 45%), or stroke
* Estimated Glomerular Filtration Rate (eGFR) < 30
* Glutamic oxaloacetic transaminase (GOT) and glutamic pyruvic transaminase (GPT) values higher than 80 U/L
* Patient with severe diabetes mellitus (HbA1C > 8%)
* Patient with alcohol addiction
* Patient with drug abuse
* Patient with infections or skin disease on the ischemic leg.
* Allergic to HA
* Patient whose blockage region only occurred in the femoral artery or at foot.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
Ankle Brachial Index (ABI) | Day 0, Week 4, Week 12, Week 24
  The percentage change of ABI from 3 follow-ups with the baseline.

SECONDARY OUTCOMES:
Clinical status (Rutherford category) | Day 0, Week 1, Week 2, Week 4, Week 12, Week 24
  Improvement in Rutherford scale was recorded at baseline and each follow-up.
Level of pain at rest | Day 0, Week 1, Week 2, Week 4, Week 12, Week 24
  Rest pain was measured using Wong-Baker FACES pain rating scale at baseline and each follow-up visit.
Ulcer size in cm2 | Day 0, Week 1, Week 2, Week 4, Week 12, Week 24
  Ulcer size was assessed and measured at each follow-up interval and compared to baseline.
Ulcer category | Day 0, Week 1, Week 2, Week 4, Week 12, Week 24
  Ulcer status was assessed at each follow-up interval and compared to baseline.
PWT/PFWT in seconds | Day 0, Week 4, Week 12, Week 24
  Peak walking time and pain-free walking time was measured at baseline and compared to W4, W12 and W24 by treadmill walking tests.
Amputation free | Week 1, Week 2, Week 4, Week 12, Week 24
  Time to below the knee amputation of the ipsilateral leg after the treatment.
Ejection fraction | Week 12, Week 24
  Ejection fraction was measured by echocardiogram to record the cardiac function at W12 and W24.
CT angiography | Week 12, Week 24
  CT angiography was performed to record the morphology of blood vessel, location, and the vessel cross section percentage.
Biochemistry | Week 12, Week 24
  Biochemistry tests were performed to interpret the health assessment at W12 and W24.
Hematology | Week 12, Week 24
  Hematology tests were performed to interpret the health assessment at W12 and W24.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No